CLINICAL TRIAL: NCT01268215
Title: The Effect of Endotracheal Instillation of Surfactant With and Without Budesonide on the Development of Bronchopulmonary Dysplasia in Ventilator-dependent, Extremely Low Birth Weight Infants: A Pilot Study
Brief Title: Pilot Study of Topical Steroid for Prevention of Chronic Lung Disease in Extremely Premature Infants.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: East Carolina University (Other)
Responsible Party: Waleed Mohammed Maamoun, MD, Neonatology Section, Pediatric Department, Brody School of Medicine at East Carolina University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UMCIRB # 10-0250
Record Dates: First submitted 2010-12-28; First posted 2010-12-29 (Estimated); Last update posted 2010-12-29 (Estimated); Status verified 2010-07

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Bronchopulmonary Dysplasia; Budesonide; Infasurf
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — calfactant; Budesonide; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (two study drugs group) (Experimental): The standard management + two study drugs (endotracheal instillation of a mixture containing budesonide and Infasurf)
  Interventions: Drug: Infasurf; Drug: Pulmicort
- B (one study drug group) (Active Comparator): The standard management + one study drug (endotracheal instillation of Infasurf only).
  Interventions: Drug: Infasurf
- C (no study drug group) (Sham Comparator): The standard management only.
  Interventions: Other: Sham

INTERVENTIONS:
Drug: Infasurf — Endotracheal instillation of Infasurf once per week for three weeks
  Other Names: Calfactant
  Arms: A (two study drugs group); B (one study drug group)
Drug: Pulmicort — Endotracheal instillation, once per week for three weeks
  Other Names: Budesonide
  Arms: A (two study drugs group)
Other: Sham — None instilled through the endotracheal tube
  Other Names: Air Sham
  Arms: C (no study drug group)

SUMMARY:
A Pilot study to evaluate the safety and the efficacy of endotracheal instillation of pulmonary surfactant, with or without topical steroid (Budesonide), as a prophylactic treatment for Bronchopulmonary Dysplasia (a form of chronic lung disease) in extremely low birth weight infants. Cytokines (a group of inflammatory mediators) are measured in the tracheal aspirate before and after instillation of the study drugs.

DETAILED DESCRIPTION:
Bronchopulmonary Dysplasia (BPD) is still one of the most common complications of ventilated premature infants. Lung inflammation plays a major role in its pathogenesis. Systemic steroids can be given to control this inflammatory process but their widespread use is limited by their systemic side effects and concerns for long neurodevelopmental adverse sequelae. Delivering steroids by inhalation which has been proven to be effective in young infants with asthma has been shown to be unsatisfactory for ELBW infants with BPD. This may be due to the fact that current delivery devices do not meet the requirements of the specific anatomical and physiologic characteristics of the airways and breathing patterns in this special group of patients. A novel approach to facilitate delivery directly to the lungs, thereby avoiding systemic concerns has been demonstrated in a recent study in which budesonide ( a topical steroid) was given to ventilated preterm infants using surfactant as a vehicle.

ELIGIBILITY:
Inclusion Criteria:

1. Birth weight 501-1000 g and ≤ 28 weeks gestational age
2. Diagnosed as RDS requiring mechanical ventilation and surfactant therapy during the first 4 hours after birth
3. Still ventilated on day 5-9 of life.
4. An interval of at least 24 hours' duration between the last dose of indomethacin and the endotracheal instillation of study drug.

Exclusion Criteria:

1. Congenital or chromosomal anomalies
2. Occurrence of perinatal sepsis
3. Use of intravenous steroids > 7 days

Ages: 24 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-06 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
To measure the effect of surfactant with and without Budesonide on the development of BPD in ELBW infants. | Supplemental oxygen requirement at 36 weeks' postmenstrual age (PMA)
  The main goal of the study is to determine whether endotracheal instillation of surfactant (Infasurf) with or without potent topical steroid (Budesonide) reduces the development of Bronchopulmonary Dysplasia (BPD) in Extremely Low Birth Weight (ELBW) infants at high risk of BPD.

SECONDARY OUTCOMES:
To measure the effect of surfactant with and without Budesonide on the inflammatory cytokines in tracheal aspirates. | The measurement of cytokines in tracheal aspirate samples will be done at the end of the study.
  Tracheal aspirate samples will be collected before instillation of each dose of the study drug, 7 days after the last dose if the infant is still intubated, and prior to elective extubation regardless of when extubation occurs. Tracheal aspirate samples will be obtained from the control (standard management) group in the same way and using the same time frame as the treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Waleed M Maamoun, MD, Principal Investigator — Pitt County Memorial Hospital/Brody School of Medicine at East Carolina University; James Cummings, MD, Study Director — Pitt County Memorial Hospital/Brody School of Medicine at East Carolina University; Scott MacGilvray, MD, Study Chair — Pitt County Memorial Hospital/Brody School of Medicine at East Carolina University; Karl Kaminski, RRT-NPS, Study Chair — Pitt County Memorial Hospital/Brody School of Medicine at East Carolina University
Locations (1):
- NICU-Pitt County Memorial Hospital, Greenville, North Carolina, United States